CLINICAL TRIAL: NCT01953354
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study of Trichuris Suis Ova Treatment in Left-sided Ulcerative Colitis and Its Effects on Mucosal Immune State and Microbiota
Brief Title: Trichuris Suis Ova Treatment in Left-sided Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: MFR's business decision to d/c TSO production -unrelated to any safety concern.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Coronado Biosciences, Inc. (Industry); Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT AUC02
Record Dates: First submitted 2013-09-24; First posted 2013-10-01 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative colitis (UC); Inflammatory Bowel Disease (IBD); Trichuris suis ova (TSO)
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trichuris suis ova (TSO) (Experimental): Six doses of TSO orally over a ten-week period
  Interventions: Biological: Trichuris suis ova (TSO)
- Placebo (Placebo Comparator): Six doses of TSO placebo orally over a ten-week period
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Trichuris suis ova (TSO) — Six doses of TSO orally over a ten-week period (e.g., every 2 weeks x 10 weeks for a total of 6 total doses)
  Other Names: T. suis ova; 7500 Trichuris suis ova (7500 TSO ); CNDO 201
  Arms: Trichuris suis ova (TSO)
Biological: Placebo — Six doses of TSO placebo orally over a ten-week period (e.g., every 2 weeks x 10 weeks for a total of 6 total doses)
  Other Names: Trichuris suis ova (TSO) placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of trichuris suis ova (TSO) in ulcerative colitis (UC). We will look at how TSO affects the body's immune response and if there are related changes in participants' UC.

DETAILED DESCRIPTION:
The cause of UC, an inflammatory bowel disease (IBD), is not well understood. It is believed to be caused from an abnormal immune response to the normal bacteria that live in the gut (intestines and colon). This response acts as an "attack" on the healthy tissue of the bowel by a person's own immune cells which leads to disease.

It is well known that autoimmune diseases such as IBD, asthma, diabetes, and multiple sclerosis are more common in industrialized, well-developed countries with better sanitation and hygiene, as in the United States. These "cleaner" environments reduce exposure to germs and parasites naturally found in the environment. This reduced exposure may trigger responses in the body that make people more prone to diseases such as UC. People in non-industrialized countries and the tropics, where parasites are common, rarely develop these diseases. This observation has led researchers to want to better understand the relationship between the lack of natural bacteria in the gut and the onset of autoimmune diseases like as UC.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. Diagnosis of UC (newly diagnosed or established patients) as determined by medical history, endoscopic and histological confirmation with the proximal disease extent limited to the left colon (distal to the splenic flexure), and accessible by flexible sigmoidoscopy. Patients with left-sided disease and the presence of a periappendiceal red patch (limited cecal inflammation) will be eligible as long as there is no intervening evidence of colitis between the cecal base and the upper boundary of inflammation in the left colon.
3. Mayo score >/= 4, as scored at Screen 2
4. If taking the following medications at Screen 1, subjects must meet the following criteria:

   1. Oral Corticosteroids: stable treatment for at least 4 weeks prior to Day 0 with a maximum dose equivalent to <\=15 mg/day of prednisone
   2. Immunosuppressants (azathioprine (AZA) or 6-mercaptopurine (6-MP)): treatment for at least 12 weeks with a stable dose, not exceeding 2.5 mg/kg/day of AZA or 1.5 mg/kg/day of 6-MP, during the 4 weeks prior to Day 0
   3. Aminosalicylates: stable oral doses up to 4.8 g/day for at least 4 weeks prior to Day 0.

Exclusion Criteria:

1. Subjects whose UC is anticipated to require surgical, endoscopic, or radiologic intervention during study participation
2. Uncontrolled GI bleeding
3. Subjects who have disease limited to the rectum (maximum disease extent of less than 15 cm)
4. Women who are pregnant, breast-feeding, or planning to become pregnant during the study. All women of childbearing potential must have a negative serum pregnancy test at Screen 2 prior to randomization of treatment.
5. Women of childbearing potential not using adequate birth control measures (e.g., total abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, surgical sterilization, Depo-Provera, or hormonal implants).
6. Current or recent serious systemic disorder including clinically significant impairment in cardiac, pulmonary, liver, renal, endocrine, hematologic, or neurologic function, based on investigator discretion
7. Subjects currently receiving the following concomitant medications:

   1. Prednisone or its equivalent at unstable doses or at doses exceeding 15 mg/day within 4 weeks prior to Day 0
   2. Local steroids such as budesonide, Colifoam, or Predsol enemas within 2 weeks prior to Screen 2
   3. Topical therapies, either mesalamine or steroids, taken within 2 weeks of Screen 2
   4. Non-steroidal anti-inflammatory drugs (NSAIDs), Cyclooxygenase (COX)-2 inhibitors, or aspirin >100 mg/day within 2 weeks prior to Screen 2
   5. Tumor necrosis factor (TNF)-alpha inhibitors including but not limited to infliximab (Remicade) or adalimumab (Humira) within 12 weeks of Day 0
   6. Any biological agent within 12 weeks of Day 0
   7. Metronidazole within 4 weeks of Day 0
   8. Receipt of any investigational agent within the 12 weeks prior to Day 0
   9. Antibacterial or oral antifungal agents within 4 weeks of Screen 2
   10. Interferon (IFN) therapy
   11. Anticoagulants
   12. Methotrexate
8. Blood transfusion within the 12 weeks prior to Day 0
9. Presence of any of the following abnormal laboratory parameters at Screen 1:

   1. Hemoglobin < 10.0 g/dL
   2. White Blood Count (WBC) < 4,000 or > 20,000/L (equivalent to WBC < 4 or > 20 x109/L)
   3. Platelets < 100,000 or > 800,000/L (equivalent to platelets < 100 or > 800 x109/L)
   4. Total bilirubin > 1.5 × Upper limit of normal (ULN)
   5. Alanine transaminase (ALT) > 2 × ULN
   6. Aspartate transaminase (AST) > 2 × ULN
   7. Alkaline phosphatase (ALK) > 1.5 × ULN
   8. Gamma-glutamyl transferase (GGT) > 1.5 × ULN
   9. Creatinine > 1.5 × ULN
10. History of drug or alcohol abuse within one year prior to Day 0
11. Inability to understand the nature and requirements of the study, or to comply with the study procedures or planned schedule of study visits
12. Evidence of infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
13. Active infection with C. difficile, bacterial enteric pathogens, or pathogenic ova/parasites
14. History of malignancy within the last 5 years, except for resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ cervical cancer Grade I
15. History of colonic dysplasia
16. Any social or medical condition that, in the opinion of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hanauer, MD, Study Chair — Northwestern University; Bana Jabri, MD, PhD, Study Chair — University of Chicago
Locations (17):
- United States (17):
  - Stanford University School of Medicine, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Summers RW, Elliott DE, Qadir K, Urban JF Jr, Thompson R, Weinstock JV. Trichuris suis seems to be safe and possibly effective in the treatment of inflammatory bowel disease. Am J Gastroenterol. 2003 Sep;98(9):2034-41. doi: 10.1111/j.1572-0241.2003.07660.x. PMID 14499784
- [Background] Moreels TG, Pelckmans PA. Gastrointestinal parasites: potential therapy for refractory inflammatory bowel diseases. Inflamm Bowel Dis. 2005 Feb;11(2):178-84. doi: 10.1097/00054725-200502000-00012. PMID 15677912
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of all the participating sites, nine reached the study intervention randomization phase for >=one participant.The first site was activated in November 2013 and the last participant was randomized in March 2015.
Groups:
- TSO 7500: Participants were randomized to receive six doses of 7500 viable, embryonated Trichuris suis ova (TSO) in liquid suspension orally over a 10-week period.
- Placebo: Participants were randomized to receive six doses of placebo in liquid suspension orally over a 10-week period.
Period: Overall Study
Arm/Group | TSO 7500 | Placebo
Started | 9 | 7
Completed | 8 | 5
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Decision of Sponsor | 0 | 1
Not completed — Disease Exacerbation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized population included all subjects who were randomized to receive either TSO 7500 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | TSO 7500 | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (9.0) | 44.7 (11.4) | 42.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16
Percentage of Participants at Baseline Who Were Taking a Corticosteroid [Number; unit: percentage of participants] — Percentage of participants at Baseline who were taking a corticosteroid prescribed by a physician.
  percentage of participants | 33.3 | 14.3 | 25.0
Percentage of Participants at Baseline Who Were Taking Thiopurine [Number; unit: percentage of participants] — Percentage of participants at Baseline who were taking Thiopurine prescribed by a physician.
  percentage of participants | 11.1 | 0.0 | 6.3
Mayo Score for Assessment of Ulcerative Colitis Activity [Mean (Standard Deviation); unit: Total Mayo Score] — The Mayo Score assesses four areas of ulcerative colitis activity: stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment. The physician rates each of the four areas on a scale of 0 to 3, with a total possible score of 12. A higher score indicates more disease activity.
  Total Mayo Score | 9.0 (1.2) | 7.4 (1.3) | 8.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Clinical Response at Week 12
Description: Clinical response is defined as a reduction in the Mayo score of at least 3 points and at least a 30% reduction from Baseline, along with either a decrease from Baseline in the rectal bleeding subscore of more than 1 point or a rectal bleeding subscore of 0 or 1.
Time Frame: Week 12
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who received at least one dose of either TSO or placebo. Only mITT subjects with clinical response results at Week 12 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 7 | 6
percentage of participants | 57.1 | 50.0
Statistical Analysis 1: Comparison: TSO 7500 vs Placebo; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

2. Secondary Outcome: Percent of Participants Who Achieved Remission at Week 12
Description: Remission is defined as a Mayo score of less than or equal to 1 with absence of rectal bleeding and endoscopy score of 0 or 1.
Time Frame: Week 12
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who received at least one dose of either TSO or placebo. Only mITT subjects with remission results at Week 12 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 7 | 6
percentage of participants | 14.3 | 16.7
Statistical Analysis 1: Comparison: TSO 7500; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

3. Secondary Outcome: Percent of Participants With Healed Colonic Mucosa at Week 12
Description: Healed colonic mucosa is defined as a Mayo endoscopy score of 0 or 1.
Time Frame: Week 12
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who received at least one dose of either TSO or placebo. Only mITT subjects with a Mayo endoscopy score at Week 12 are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 6 | 6
percentage of participants | 66.7 | 16.7
Statistical Analysis 1: Comparison: TSO 7500 vs Placebo; Test type: Superiority or Other; p = 0.242, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

4. Secondary Outcome: Percent of Participants With a Modified Clinical Response
Description: Modified clinical response is defined as a reduction in the modified Mayo score (i.e., minus the endoscopy component) of at least 2 points from baseline.
Time Frame: From Day 0 through time of first clinical response or end of follow-up, whichever comes first, up to 12 Weeks
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who received at least one dose of either TSO or placebo. Only mITT subjects with baseline and at least one post-baseline modified clinical response result are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 9 | 7
percentage of participants | 88.9 | 71.4
Statistical Analysis 1: Comparison: TSO 7500 vs Placebo; Test type: Superiority or Other; p = 0.550, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

5. Secondary Outcome: Time to Modified Clinical Response
Description: Number of days to reach a modified clinical response. Modified clinical response is defined as a reduction in the modified Mayo score (i.e., minus the endoscopy component) of at least 2 points from baseline.
Time Frame: From Baseline through the day that modified clinical response is reached. Week 16 is the last visit that the modified Mayo score is assessed.
Population: The Modified Intent-to-Treat (mITT) population included all randomized subjects who received at least one dose of either TSO or placebo. Only mITT subjects who achieved a modified clinical response are included in this analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 8 | 5
Days | 34.5 [14 to 125] | 28.0 [15 to 126]

6. Secondary Outcome: Percent of Participants With Colonoscopic Evidence of Visible Worm
Description: Stool evaluations for ova and parasites confirmed the absence of T. suis. If evidence suggested a presence of T. suis, a colonoscopy would be performed to confirm invasion with a visible worm.
Time Frame: From Day 0 through end of follow-up, up to 36 weeks
Population: The Safety population included all subjects for whom study treatment was initiated.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 9 | 7
percentage of participants | 0 | 0

7. Secondary Outcome: Percent of Participants With Increase in Diarrhea
Description: An increase in diarrhea is defined as an increase in the Mayo Score's Stool Frequency score by at least 1 point from baseline at any time during follow-up.
Time Frame: From Day 0 through end of follow-up, up to 36 weeks
Population: The Safety population included all subjects for whom study treatment was initiated.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 9 | 7
percentage of participants | 11.1 | 28.6
Statistical Analysis 1: Comparison: TSO 7500 vs Placebo; Test type: Superiority or Other; p = 0.550, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

8. Secondary Outcome: Percent of Participants With Increase in Concurrent Ulcerative Colitis (UC) Medications or New Rescue Medications Added
Description: New or increase in UC medications is defined as a need for dose-escalation of concurrent medications or need for rescue medications to treat UC through Week 16.
Time Frame: From Day 0 through Week 16
Population: The Safety population included all subjects for whom study treatment was initiated.
Measure: Number; unit: percentage of participants
Arm/Group | TSO 7500 | Placebo
Number analyzed (Participants) | 9 | 7
percentage of participants | 44.4 | 28.6
Statistical Analysis 1: Comparison: TSO 7500 vs Placebo; Test type: Superiority or Other; p = 0.633, Fisher Exact — P-value is testing for a difference in proportions using a Fisher's exact test

ADVERSE EVENTS:
Time Frame: From the time of signed informed consent to the required follow-up time (Week 36) or until 30 days after the participant prematurely withdrew from the study.
Description: CTCAE V4.0
Arm/Group | TSO 7500 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/8 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSO 7500 (N=8) | Placebo (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was slower than anticipated. The study was ultimately terminated when the manufacturer decided to discontinue study product production.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No